CLINICAL TRIAL: NCT04908696
Title: Department of Otorhinolaryngology, Eye & ENT Hospital
Brief Title: Clinical Treatments in Specialized Diseases of Laryngeal Carcinoma (LC) and Hypopharyngeal Carcinoma (HPC)
Status: Recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Changhai Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Fudan University (Other); Shanghai Changzheng Hospital (Other); RenJi Hospital (Other); Shanghai 6th People's Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, LeiTao, Director, Eye & ENT Hospital of Fudan University
Other Study IDs: LC & HPC T121
Record Dates: First submitted 2021-05-24; First posted 2021-06-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Glottic Carcinoma; Supraglottic Carcinoma; Subglottic Carcinoma; Pyriform Sinus Carcinoma; Postcricoid Carcinoma; Posterior Pharyngeal Wall Carcinoma
Keywords: Laryngeal carcinoma; Hypopharyngeal carcinoma; Surgery; Laryngeal function preservation treatment
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — Radiotherapy; Chemoradiotherapy; Neoadjuvant Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- TLM treatment for LC and PHC patients with early stage: TLM group: Laryngeal carcinoma (LC) (supraglottic type and glottic type) and hypopharyngeal carcinoma (HPC) (pyriform sinus and posterior pharyngeal wall) patients with T1 and T2 stages can be treated with transoral laser microsurgery (CO2 laser resection) for proper indications (NCCN 2020).
  Interventions: Procedure: routines
- OPL treatment for LC and PHC patients with T1, T2, and T3 stages: OPL group: Open partial laryngectomy with laryngeal function preservation is performed for patients with laryngeal carcinoma (LC) (supraglottic type, glottic type, and subglottic type) and hypopharyngeal carcinoma (PHC) (pyriform sinus, postcricoid, and posterior pharyngeal wall) with proper indications (NCCN 2020).
  Interventions: Procedure: routines
- R treatment for LC and PHC patients with early stage: R group: radiotherapy is treated for laryngeal carcinoma (LC) and hypopharyngeal carcinoma (PHC) patients with early stage with proper indications (NCCN 2020).
  Interventions: Procedure: routines
- TORS treatment for LC and PHC patients with early stage: TORS group: transoral robotic surgery is performed for proper laryngeal carcinoma (LC) and hypopharyngeal carcinoma (PHC) patients with early stage with proper indications.
  Interventions: Procedure: routines
- SPA treatment for LC and PHC patients with advanced stage: SPA group: surgical treatment (S) ± postoperative adjuvant (PA) therapy is performed for laryngeal carcinoma (LC) and hypopharyngeal carcinoma (PHC) patients with advanced stage with proper indications (NCCN 2020).
  Interventions: Procedure: routines
- CCR treatment for LC and PHC patients with advanced stage: CCR group: concurrent chemoradiotherapy (CCR) is performed for laryngeal carcinoma (LC) and hypopharyngeal carcinoma (PHC) patients with advanced stage with proper indications (NCCN 2020).
  Interventions: Procedure: routines
- ARC treatment for LC and PHC patients with advanced stage: ARC group: neoadjuvant therapy (A) + radiotherapy/chemoradiotherapy (RC) is performed for laryngeal carcinoma (LC) and hypopharyngeal carcinoma (PHC) patients with advanced stage with proper indications (NCCN 2020).
  Interventions: Procedure: routines
- ASRC treatment for LC and PHC patients with advanced stage: ASRC group: neoadjuvant therapy (A) + surgery (S) + radiotherapy (R) or chemoradiotherapy (C) is performed for laryngeal carcinoma (LC) and hypopharyngeal carcinoma (PHC) patients with advanced stage with proper indications (NCCN 2020).
  Interventions: Procedure: routines

INTERVENTIONS:
Procedure: routines — For early stage laryngeal carcinoma and hypohparyngeal carcinoma (T1 and T2), transoral laser microsurgery (CO2 laser resection), open partial laryngectomy (vertical partial laryngectomy, cricohyoidoepiglottopexy, cricohyoidopexy, horizontal partial laryngectomy), partial hypopharyngectomy, radiotherapy, and transoral robotic surgery were performed for patients with proper indications (NCCN 2020).
  For advanced stage laryngeal carcinoma and hypohparyngeal carcinoma (T3 and T4), surgical treatment ± postoperative adjuvant therapy, concurrent chemoradiotherapy, neoadjuvant therapy + radiotherapy/chemoradiotherapy, or neoadjuvant therapy + surgery + radiotherapy or chemoradiotherapy were performed for patients with proper indications (NCCN 2020).
  Other Names: Open partial laryngectomy with laryngeal function preservation; Radiotherapy; Transoral robotic surgery; Surgical treatment ± postoperative adjuvant therapy; Concurrent chemoradiotherapy; Neoadjuvant therapy + radiotherapy/chemoradiotherapy; Neoadjuvant therapy + surgery + radiotherapy or chemoradiotherapy

SUMMARY:
For early stage laryngeal carcinoma and hypohparyngeal carcinoma (T1 and T2), transoral laser microsurgery, open partial laryngectomy, radiotherapy, and transoral robotic surgery were performed according to NCCN guidelines (2020).

For advanced stage laryngeal carcinoma and hypohparyngeal carcinoma (T3 and T4), surgical treatment ± postoperative adjuvant therapy, chemoradiotherapy, neoadjuvant therapy + radiotherapy/chemoradiotherapy, or neoadjuvant therapy + surgery + radiotherapy or chemoradiotherapy performed according to NCCN guidelines (2020).

This study plan to analyze the clinical ouctomes of different treatment for the same T stage disease. The overall survival rate, disease specific survival, disease free survival, local control, regional control, and laryngeal function preservation rate were analyzed in this study.

DETAILED DESCRIPTION:
For early stage laryngeal carcinoma and hypohparyngeal carcinoma (T1 and T2), transoral laser microsurgery (CO2 laser resection), open partial laryngectomy (vertical partial laryngectomy, cricohyoidoepiglottopexy, cricohyoidopexy, horizontal partial laryngectomy), partial hypopharyngectomy, radiotherapy, and transoral robotic surgery were performed for patients with proper indications.

For advanced stage laryngeal carcinoma and hypohparyngeal carcinoma (T3 and T4), surgical treatment ± postoperative adjuvant therapy, concurrent chemoradiotherapy, neoadjuvant therapy + radiotherapy/chemoradiotherapy, or neoadjuvant therapy + surgery + radiotherapy or chemoradiotherapy were performed for patients with proper indications.

This study seek to analyze and compare the clinical ouctomes of different treatments for the same T stage disease of LC and HPC.

The main end events involving overall survival rate, disease specific survival rate, and laryngeal function preservation rate were analyzed in this study. Beside, the events of disease free survival rate, local control rate, and regional control rate were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Laryngeal cancer: glottic type, supraglottic type, and subglottic type; hypopharyngeal cancer: pyriform sinus type, postcri-coid type, and posterior pharyngeal wall type.
* T1, T2, T3, and T4 stage.
* Age 18 - 90.
* Male or female.
* Good compliance.
* No other severe related diseases that may impact the treatment (such as other tumors, severe heart, lung and central nervous system diseases, etc.).
* Negative pregnancy test (for female patients with fertility).
* Male patients with fertility and female patients with fertility and pregnancy risk must agree to use contraceptive methods throughout the study period, and continued until at least 6 months after the last dose of cisplatin. Female patients do not have fertility. Female patients with postmenopausal status.

Exclusion Criteria:

* Patients who have previously been diagnosed with immunodeficiency or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related diseases.
* Patients with a known history of active tuberculosis (TB).
* Pregnant women or lactating women.
* The doctors believes that it is inappropriate for patients to participate in the trial: having, for example, severe acute or chronic medical conditions (including immune colitis, inflammatory bowel disease, non-infectious pneumonia, pulmonary fibrosis) or mental illness (including recent time [within the past year] or active suicidal ideation or behavior).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort study involve laryngeal cancer and hypopharyngeal cancer patients with T1 -T4 stages, and we plan to observe the oncologic outcomes from different clinical treatments.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-23 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
3 - years overall survival | Three years
  the time between the treatment and the date of death from any causes
3 - years disease specific survival | Three years
  the time between the treatment and the date of death from laryngeal carcinoma or hypohparyngeal carcinoma
3 - years laryngeal function preservation | Three years
  the time between the treatment and the date of laryngeal function preservation failure

SECONDARY OUTCOMES:
3 - years disease free survival | Three years
  the time between the treatment and the first evidence of disease recurrence, metastasis or death
3- local control | Three years
  the time between the treatment and the first evidence of local recurrence
3- regional control | Three years
  the time between the treatment and the first evidence of regional recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Lei Tao, Dr., Study Chair — Department of Otorhinolaryngology, Eye & ENT Hospital, Fudan University, Shanghai, China
Locations (1):
- Lei Tao, Shanghai, Shanghai Municipality, China